CLINICAL TRIAL: NCT00582517
Title: Compass Hinge Stabilization of Knee Dislocations: A Randomized Trial
Acronym: CKH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Theiss, MD, Study Coordinator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F000330008; OGCA Contract #200497 (Other: UAB Link Number)
Record Dates: First submitted 2007-12-18; First posted 2007-12-28 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Knee Dislocation
Keywords: Orthopaedic Trauma; Knee Dislocation; Compass Hinge External Fixator; External Brace
MeSH Terms: conditions — Knee Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A External Brace (Active Comparator): Group A will have a non-invasive range of motion external brace placed following surgery
  Interventions: Procedure: Non-invasive External Knee Brace
- Group B Compass Knee Hinge (Experimental): Group B will have a Compass Knee Hinge placed
  Interventions: Device: Compass Universal Hinge External Fixator

INTERVENTIONS:
Device: Compass Universal Hinge External Fixator — Application of the Compass Knee Hinge adds approximately 30 minutes to the surgical time. After the apparatus has been in place for the appropriate amount of time (6-8 weeks), it is removed either in the clinical setting, or in the one-day surgery area of UAB Highlands.
  Other Names: Compass Knee Hinge
  Arms: Group B Compass Knee Hinge
Procedure: Non-invasive External Knee Brace — For Group A patients, an external knee brace (several brands available and no one brace specified for this study) will be placed on the leg following surgical repair of the knee dislocation.
  Arms: Group A External Brace

SUMMARY:
The purpose of this project is to evaluate the effect of the Compass™ Universal Hinge external fixator on the outcome of patients following acute dislocation of the knee

DETAILED DESCRIPTION:
Prospective randomized outcome study. Patients will be randomized either into the control group (Group A) or the study group (Group B) based on a computer generated randomization table. Both groups will undergo an identical surgical protocol, as outlined below. The only difference is that patients in Group A will have a range of motion external brace placed following surgery, while patients in Group B will have a CKH placed. The rehabilitation protocol for the two groups will be identical, as outlined below. Both groups will undergo an Anterior Cruciate Ligament (ACL) reconstruction on a delayed basis two months following surgery, if the ACL was torn during the knee dislocation. The ACL reconstruction will be delayed in both groups if a minimum range of motion of 10-90 degrees has not been attained.

Surgical Protocol : Approximately 10 - 21 days following the injury, patients will undergo the first surgical procedure on their knee dislocation. During the first procedure, they will have a Posterior Cruciate Ligament (PCL) reconstruction using an achilles tendon allograft, with the direct onlay, two bundle technique. Additionally, any damage to either the posterior medial or posterior lateral corner will be repaired (not reconstructed), and any meniscus pathology will be addressed. The final step of this first procedure will be applying the CKH to patients randomized to the compass group (the alignment pins will be placed prior to repair of the corner). Patients will undergo an ACL reconstruction (if necessary) approximately 8 weeks following the initial surgery, when the CKH will be removed. Additional surgeries will be performed on patients to treat motion problems/arthrofibrosis as well as recurrent instability on an "as-needed basis."

Rehabilitation Protocol - aggressive rehabilitation will be started on the day following surgery. Patients will be placed in Continuous Passive Motion (CPM) machines with an initial range of motion of 0 - 30 degrees. The hinge will be locked into full extension for at least 4 hours per day. We will continue CPM for two weeks, with a goal of increasing by at least 10 degrees per day to 90 degrees of flexion. Weightbearing will be allowed as tolerated with the hinge locked in extension.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient with a knee dislocation that requires surgical repair
* Adult patient (19 years and older)

Exclusion Criteria:

* Patients unable or unwilling to comply with follow-up gait, radiographic and clinical evaluations necessary to complete the study
* Patients unable or unwilling to give informed consent and/or who have no responsible family member willing to give consent
* Pregnant women
* Prisoners

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Volgas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Result] Stannard JP, Sheils TM, McGwin G, Volgas DA, Alonso JE. Use of a hinged external knee fixator after surgery for knee dislocation. Arthroscopy. 2003 Jul-Aug;19(6):626-31. doi: 10.1016/s0749-8063(03)00125-7. PMID 12861201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A External Brace | Group B Compass Knee Hinge
Started | 45 | 55
Completed | 45 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A External Brace | Group B Compass Knee Hinge | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 52 | 97
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 37 | 39 | 76
Region of Enrollment [Number; unit: participants]
  United States | 45 | 55 | 100

OUTCOME MEASURES:

1. Primary Outcome: Knee Stability
Description: The hypothesis of this study was that there would be equivalent final knee range of motion with fewer failures for ligament reconstructions following knee dislocations that were supplemented with the Compass Knee Hinge as compared to a control group.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Group A External Brace: Group A will have a non-invasive range of motion external brace placed following surgery. Stability of the knee determined by Continuous Passive Motion (CPM) machines and range of motion reached.
- Group B Compass Knee Hinge: Group B will have a Compass Knee Hinge placed. Stability of the knee determined by Continuous Passive Motion (CPM) machines and range of motion reached.
Arm/Group | Group A External Brace | Group B Compass Knee Hinge
Number analyzed (Participants) | 45 | 55
participants
  Stable at 30 degree plane | 29 | 26
  Unstable at 30 degree plane | 12 | 17
  Stable at 70 degree plane | 27 | 30
  Unstable at 70 degree plane | 14 | 13
  Stable at 90 degree plane | 4 | 12

ADVERSE EVENTS:
Time Frame: Baseline to 12 months
Arm/Group | Group A External Brace | Group B Compass Knee Hinge
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 0/45 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No